CLINICAL TRIAL: NCT04512248
Title: Integrating the Quit and Stay Quit Monday Model Into Smoking Cessation Services for Smokers With Mental Health Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 20-01247
Record Dates: First submitted 2020-08-11; First posted 2020-08-13 (Actual); Last update posted 2022-01-05 (Actual); Status verified 2021-12

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Intervention Model Description: Two-group, parallel-randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Quit and Stay Quit Monday Model (Experimental)
  Interventions: Behavioral: Quit and Stay Quit Monday Model
- Usual Care (No Intervention)

INTERVENTIONS:
Behavioral: Quit and Stay Quit Monday Model — Participants randomized to the study intervention will receive: (1) 2 telephone smoking cessation coaching calls; (2) enrollment into SmokefreeTXT; and (3) enrollment in the iquitmonday.org weekly email newsletter. The telephone coaches will ask these participants to identify a future Monday as their quit date and provide coaching to achieve a Monday quit. The coaches will also enter the selected Monday as the patient's quit day when enrolling the patient into SmokefreeTXT.
  Arms: Quit and Stay Quit Monday Model

SUMMARY:
The Quit and Stay Quit Monday model is an innovative smoking cessation approach that guides smokers' behavior without requiring additional resources. The investigator will conduct a randomized control trial evaluating the effectiveness of this model as compared to usual smoking cessation care in a population of smokers with a mental health condition.

DETAILED DESCRIPTION:
The overall objective of this proposal is to innovate the tobacco treatment paradigm for smokers with mental health conditions (MHC) by integrating the Quit and Stay Quit Monday Model into smoking cessation services for this vulnerable population.

The investigator will conduct a two-group, parallel-randomized controlled trial (RCT). The target population will be generated by the NYU Langone electronic medical record (EMR). The investigator will proactively contact patients to offer enrollment and randomize participants 1:1 to one of two groups (n=50/group): (1) Quit and Stay Quit Monday Model or (2) Usual Care. For evaluation, phone surveys will be conducted at baseline and 3-months to assess quit attempts, intervention satisfaction, and smoking cessation.

ELIGIBILITY:
Inclusion Criteria:

1. age ≥ 18 years old
2. Has smoked a cigarette in the past 30 days, even a puff
3. Has been diagnosed with a mental health condition or received care from a mental health clinic within the NYU Langone Health system in the prior 12 months
4. Interested in quitting smoking
5. English language
6. Has a phone that can receive text messages
7. Able to provide informed consent

Exclusion Criteria:

1. age < 18 years of age
2. Non-smoker

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-10-30 (Actual); Study Completion 2021-10-30 (Actual)

PRIMARY OUTCOMES:
Incidence of 3-month quit attempts | 3 months
  Phone surveys will be conducted to obtain information
Incidence of smoking cessation | 3 months
  Phone surveys will be conducted to obtain information
Number of participants who report satisfaction in intervention | 3 months
  Phone surveys will be conducted to obtain information

CONTACTS AND LOCATIONS:
Overall Officials: Erin Rogers, DrPH, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices) will be shared upon reasonable request.
Supporting Information: Study Protocol, SAP
Time Frame: Data will become available beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will have access to the data upon reasonable request. Requests should be directed to ERIN.ROGERS@NYULANGONE.ORG. To gain access, data requestors will need to sign a data access agreement.

REFERENCES:
- [Derived] Vojjala M, Wysota CN, Oketunbi O, King Q, Rogers ES. Integrating the "Quit and Stay Quit Monday" Model into Smoking Cessation Services for Smokers with Mental Health Conditions: A Pilot Randomized Controlled Trial. J Smok Cessat. 2023 Jul 22;2023:8165232. doi: 10.1155/2023/8165232. eCollection 2023. PMID 37521160